CLINICAL TRIAL: NCT06980337
Title: Combined Effect of Kendall and Scapulothoracic Exercises on Brachial Plexus Mechanoreceptors in Chronic Non-specific Neck Pain
Brief Title: Effect of Kendall and Scapulothoracic Exercises in Treatment of Chronic Non-specific Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, Assistant professor of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Physical Therapy 52025; Faculty of Physical therapy (Other: Cairo university)
Record Dates: First submitted 2025-05-08; First posted 2025-05-20 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Non-specific Chronic Neck Pain
Keywords: chronic non-specific neck pain; Kendall exercises; Scapulothoracic exercises; Brachial Plexus mechanoreceptors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A will receive conventional treatment (Experimental)
  Interventions: Other: Conventional treatment program
- Group B will receive scapulothoracic exercises and conventional treatment. (Experimental)
  Interventions: Other: Conventional treatment program; Other: Scapulothoracic exercises
- Group C will receive Kendall exercises, scapulothoracic exercises and conventional treatment (Experimental)
  Interventions: Other: Conventional treatment program; Other: Scapulothoracic exercises; Other: Kendall exercises

INTERVENTIONS:
Other: Conventional treatment program — Ultrasound, hot packs, cervical postural stretching and strengthening exercise will be done for all groups.
  Stretching Exercises Posture correction exercises training will include stretching of tight muscles such as Pectoralis major, levator scapulae, upper trapezius, suboccipital muscles and, sternocleidomastoid.
  Strengthening Exercises Exercises will include Chin Tucks exercise and Neck isometric exercises
Other: Scapulothoracic exercises — Scapulothoracic exercises It is a strengthening exercises of the serratus anterior muscle, as well as the middle and inferior fibres of the trapezius muscle
  Arms: Group B will receive scapulothoracic exercises and conventional treatment.; Group C will receive Kendall exercises, scapulothoracic exercises and conventional treatment
Other: Kendall exercises — The exercise techniques used by Kendell were as follows:
  1. Stretching of the Cervical Extensors: By sitting with the head down and putting both hands across the occipital area, the cervical extensors can be stretched by adopting a flex neck position 2- Strengthening of the Deep Cervical Flexors Positioning supine with the chin tucked in and lifting the head for 2 to 8 s 3- Strengthening the Shoulder Retraction Maintaining an upright posture, keep the resistance band circling with strong support and stretching it with the upper limbs of both sides so that there is full retraction of the scapula 4-Stretching the Pectorals muscle Assigning both hands on the occipital area and pulling the elbows back up (bilateral) and performance arm abduction and external rotation (unilateral).
  Arms: Group C will receive Kendall exercises, scapulothoracic exercises and conventional treatment

SUMMARY:
The purpose of the clinical trial is to investigate the effect of the combined Kendall and scapulothoracic exercises program on mechanosensitivity of brachial plexus, cervical range of motion, neck functional ability, and craniovertebral angle in patients with chronic non-specific neck pain.

we have 3 groups to compare between traditional treatment, scapulothoracic and kendall exercises in treatment of chronic non-specific neck pain.

DETAILED DESCRIPTION:
Non-specific neck pain is a generalized pain in the neck and/or shoulder that has mechanical characteristics, such as symptoms brought on by holding a certain neck position, moving the neck, or palpating the cervical muscles (Fernández-de-las-Penas et al., 2007). Minor injuries to the neck caused by poor posture and abrupt muscle contractions might further cause the muscles that are not frequently utilized to shrink, which can result in mechanical dysfunction and chronic pain (Boyd-Clark et al., 2002).

Kendall exercise is generally used as physical therapy for forward head posture and induces proper neck alignment generally using strengthening methods for two muscles (deep cervical flexors and retractors of the scapula) and stretching methods for two muscles (neck extensor muscles and pectoralis) to help with forward head posture, which is a state of imbalance of muscles) (Kendall et al., 2005).

Scapulothoracic strength training may have positive impacts across subjective and objective parameters including pain, and sequentially, activities of daily living, neck range of motion, and strength (Anna-Maria et al., 2020)

PURPOSE:

The purpose of study is to investigate the effect of the combined Kendall and scapulothoracic exercises program on mechanosensitivity of brachial plexus, cervical range of motion, neck functional ability, and craniovertebral angle in patients with chronic non-specific neck pain.

* The mechanosensitivity of brachial plexus will be measured with strength duration curve
* CROM will be used to measure cervical range of motion
* Neck disability index will be used to evaluate and document neck functional ability in patients with neck pain.
* Kinovea software program will be used to measure the craniovertebral angle of the cervical spine by still photography The subjects will receive treatment for four weeks all variables wil be measured pre-treatment and post treatment

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients of both genders were recruited in the study.
* The age of the recruited subjects were ranging from 25 to 50 years old
* Patients having neck pain symptoms provoked by neck postures, neck movement, or palpation of the cervical musculature, for at least the last 3 months
* Patients with a craniovertebral angle of less than 54º
* Subjects with a BMI 25-30

Exclusion Criteria:

* History of previous injury of the neck
* History of surgical intervention at the neck
* History of inflammatory joint disease affecting facet joints
* Neurological disorders such as cervical spondylosis, spondylolisthesis or disc prolapse (Kim et al., 2012).
* Rheumatic diseases.
* Cancer patients
* Patients who received pain medication or physical therapy for their neck pain during the last 3 months
* Patients who are unable to perform the exercises.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The strength-duration curve to assess the change in mechanosensitivity of brachial plexus | at first week and after 4 weeks of treatment
  The mechanosensitivity of brachial plexus will be measured with strength duration curve by EMG. Assessment will be before and after treatment

SECONDARY OUTCOMES:
Change in Cervical range of motion | at first week and after 4 weeks of treatment
  Cervical range of motion will assessed by Cervical Range of Motion (CROM) device . Assessment will be before and after treatment
Change in Functional performance will be measured by Neck disability index | at first week and after 4 weeks of treatment
  Neck functional ability assessed by Neck disability index. Assessment will be before and after treatment
Change in Craniovertebral angle | at first week and after 4 weeks of treatment
  Craniovertebral angle assessd by Kinovea software program. Assessment will be before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Noha Elserty Assistant professor of physical therapy - Benha University, Assistant professor, Study Director — Department of Basic sciences for physical therapy, Faculty of Physical Therapy , Benha university, Benha, Egypt
Locations (1):
- Physical therapy College - Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No